CLINICAL TRIAL: NCT03590262
Title: Effect of Metformin as add-on Therapy on Glycemic Control and Other Diabetes-Related Outcomes in Type 1 Diabetic Patients:a Open-label,Self-control Study
Brief Title: Effect of Metformin as add-on Therapy on Glycemic Control and Other Outcomes in Type 1 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 723
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes Mellitus; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metformin (Experimental): patients take metformin 500mg twice or three times a day as add-on therapy to insulin for 3 months ,using self-control method.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — take the metformin 500mg twice or three times a day
  Other Names: metformin hydrochloride tablets

SUMMARY:
Aim Evidence of a possible connection between gut microbiota and several physiological processes linked to type 1 diabetes is increasing. However, the effect of multistrain probiotics in people with type 1 diabetes remains unclear. This study investigated the effect of metformin as add-on therapy on glycemic control and other diabetes-related outcomes in people with type 1 diabetes.

DETAILED DESCRIPTION:
Design An open-label, add-on, self-control clinical trial. Setting Diabetes clinic of a teaching hospital in Shenzhen China Participants A total of 20 participants with type 1 diabetes, aged 18-60 years, will be recruited and treated with metformin as add-on therapy with insulin for 12 weeks.

Outcomes Primary outcomes were glycemic control related parameters, and secondary outcomes were anthropomorphic variables, lipid profile, blood pressure and high-sensitivity C-reactive protein. The gut microbiota profile will be analyzed before and after intervention .

ELIGIBILITY:
Inclusion Criteria:

type 1 diabetes patients age 18-60years old 18 Kg/m2≤BMI≤30Kg/m2 ketonuria (-)；

Exclusion Criteria:

pregnancy lactation having other severe chronic illnesses taking other anti-diabetic drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of hemoglobin A1c in percentage | 3 months
  analyze the change of hemoglobin A1c before and after the treatment

SECONDARY OUTCOMES:
Change of weight in kilograms | 3 months
  analyze the change of weight in kilograms before and after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fengyi Yuan, Principal Investigator — associate chief physician
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided